CLINICAL TRIAL: NCT01944878
Title: Retrospective Observational Study of Impact of Portal Hypertension for the Peptic Ulcer in Liver Cirrhosis and Chronic Hepatitis
Brief Title: The Association With Peptic Ulcer Disease and Hepatic Vein Pressure Gradient
Status: Completed | Type: Observational
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Chang Seok Bang, Principal investigator, Chuncheon Sacred Heart Hospital
Other Study IDs: BCS-1
Record Dates: First submitted 2013-09-06; First posted 2013-09-18 (Estimated); Results first posted 2014-07-24 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Cirrhosis; Chronic Liver Disease
Keywords: Peptic ulcer; Liver cirrhosis; Portal hypertension
MeSH Terms: conditions — Fibrosis; Peptic Ulcer; Liver Cirrhosis; Hypertension, Portal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with chronic hepatitis: Patients with chronic hepatitis, who experienced HVPG measurement via transjugular approach and EGD within 3 months of HVPG measurement
- Patients with liver cirrhosis: Patients with liver cirrhosis, who experienced HVPG measurement via transjugular approach and EGD within 3 months of HVPG measurement

SUMMARY:
The aim of this study is to assess the role of portal hypertension of peptic ulcer disease in liver cirrhosis and chronic hepatitis.

DETAILED DESCRIPTION:
Retrospective case-control study

* Investigators will analyze the medical records of hepatic vein pressure gradient (HVPG) and esophagogastroduodenoscopy (EGD) cases who had liver cirrhosis (LC) or chronic hepatitis in a single tertiary hospital (Chuncheon Sacred Heart hospital, Korea) within 2008~2012.
* Portal hypertension is assessed using HVPG measurement via transjugular approach.
* Peptic ulcer is evaluated through EGD within 3 months of HVPG measurement
* The association of Peptic ulcer with LC, chronic hepatitis and total population (LC or chronic hepatitis) will be assessed by univariate and multivariate analysis
* There is no specific time frame, because this study is retrospective observational study, however EGD data is enrolled if it was done within 3 month from HVPG measurement.

ELIGIBILITY:
Inclusion Criteria:

* The patients who underwent hepatic vein pressure gradient (HVPG) measurement and esophagogastroduodenoscopy (EGD) and also had LC or chronic hepatitis

Exclusion Criteria:

* The patients who have missing or incomplete HVPG or EGD data
* The patients who underwent gastrectomy
* The patients who have systemic malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators will analyze the medical records of hepatic vein pressure gradient (HVPG) and esophagogastroduodenoscopy (EGD) cases who had LC or chronic hepatitis in single tertiary hospital of Korea.
Sampling Method: Non-Probability Sample
Enrollment: 455 (Actual)
Dates: Start 2013-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chang Seok Bang, M.D, Principal Investigator — Department of Internal Medicine, Hallym University College of Medicine; Gwang Ho Baik, M.D, Study Chair — Department of Internal Medicine, Hallym University College of Internal Medicine
Locations (1):
- Chuncheon Sacred Heart hospital, Chuncheon, Gangwon-do, South Korea

REFERENCES:
- [Background] Siringo S, Burroughs AK, Bolondi L, Muia A, Di Febo G, Miglioli M, Cavalli G, Barbara L. Peptic ulcer and its course in cirrhosis: an endoscopic and clinical prospective study. J Hepatol. 1995 Jun;22(6):633-41. doi: 10.1016/0168-8278(95)80219-3. PMID 7560857
- [Background] Vergara M, Calvet X, Roque M. Helicobacter pylori is a risk factor for peptic ulcer disease in cirrhotic patients. A meta-analysis. Eur J Gastroenterol Hepatol. 2002 Jul;14(7):717-22. doi: 10.1097/00042737-200207000-00002. PMID 12169979
- [Background] Kamalaporn P, Sobhonslidsuk A, Jatchavala J, Atisook K, Rattanasiri S, Pramoolsinsap C. Factors predisposing to peptic ulcer disease in asymptomatic cirrhotic patients. Aliment Pharmacol Ther. 2005 Jun 15;21(12):1459-65. doi: 10.1111/j.1365-2036.2005.02507.x. PMID 15948813
- [Derived] Bang CS, Baik GH, Kim JH, Kim JB, Suk KT, Yoon JH, Kim YS, Kim DJ. Peptic ulcer disease in liver cirrhosis and chronic hepatitis: impact of portal hypertension. Scand J Gastroenterol. 2014 Sep;49(9):1051-7. doi: 10.3109/00365521.2014.923501. Epub 2014 Jun 5. PMID 24902119

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We analyzed the medical records of 455 hepatic vein pressure gradient (HVPG) and esophagogastroduodenoscopy (EGD) patients who had LC or chronic hepatitis in a single tertiary hospital.
Pre-assignment Details: 800 HVPG measurement cases (Initial). Missing data (3), failure of HVPG measurements (8), cases without EGD (196); including 35 cases of patients on B-blocker, EGD over 3 months from HVPG measurement (79), incomplete EGD due to remnant food materials (19), cases having a history of gastrectomy (5), acute hepatopathy (5), and HCC (30) were excluded.
Period: Overall Study
Arm/Group | Patients With Chronic Hepatitis | Patients With Liver Cirrhosis
Started | 127 | 328
Completed | 127 | 328
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of 127 patients with chronic hepatitis and 328 patients with liver cirrhosis were enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients With Chronic Hepatitis | Patients With Liver Cirrhosis | Total
Number analyzed (Participants) | 127 | 328 | 455
Age, Continuous [Median (Inter-Quartile Range); unit: years] — This is the median age and interquartile range of enrolled patients divided by group (chronic hepatitis vs. liver cirrhosis)
  years | 45 [37 to 54] | 52 [46 to 59] | 50 [44 to 57]
Sex: Female, Male [Count of Participants; unit: Participants] — The number of gender distribution is described in each group here.
  Participants
    Female | 46 | 70 | 116
    Male | 81 | 258 | 339
HVPG (mmHg) [Median (Inter-Quartile Range); unit: mmHg] — HVPG (Hepatic vein pressure gradient) was measured in the enrolled population. HVPG reflects portal pressure of patient. To find the relationship between peptic ulcer disease and portal hypertension, the Fisher's exact test was performed.
  mmHg | 3.5 [2 to 5.5] | 15 [10.78 to 20] | 12 [5 to 18.3]
PUD [Number; unit: participants] — This is the number of peptic ulcer disease patients in the each group (patients with chronic hepatitis vs. patients with liver cirrhosis)
  participants | 13 | 59 | 72
Medication (NSAIDs, aspirin, clopidogrel, ticlopidine, steroid) [Number; unit: participants] — The number of patients who taking medication in each group is described here.
  participants | 7 | 16 | 23
smoking [Number; unit: participants] — The number of smokers in each group is described here.
  participants | 39 | 164 | 203
alcoholc [Number; unit: participants] — The number of alcoholics in each group is described here.
  participants | 56 | 233 | 289

OUTCOME MEASURES:

1. Primary Outcome: The Association of HVPG and PUD in Patients With Liver Cirrhosis
Description: The association of hepatic vein pressure gradient that reflects portal hypertension and peptic ulcer disease in patients with liver cirrhosis was assessed statistically.
  (NO specific time frame, only confined to 2009 to 2012, when the HVPG measurement was done). The Mann-Whitney test was used to evaluate the association between PUD or not and HVPG degree, by SPSS software.
Time Frame: Retrospective case-control study (from 2009 to 2012, up to 3 years)
Measure: Median (Inter-Quartile Range); unit: mmHg
Groups:
- PUD in Liver Cirrhosis: Patients with PUD in liver cirrhosis, who experienced HVPG measurement via transjugular approach and EGD within 3 months of HVPG measurement
- No PUD in Liver Cirrhosis: Patients without PUD in liver cirrhosis, who experienced HVPG measurement via transjugular approach and EGD within 3 months of HVPG measurement
Arm/Group | PUD in Liver Cirrhosis | No PUD in Liver Cirrhosis
Number analyzed (Participants) | 59 | 269
mmHg | 14.5 [11.5 to 19.5] | 15.3 [10.2 to 20.3]

2. Secondary Outcome: The Association Between PUD and HVPG in Patients With Chronic Hepatitis
Time Frame: Retrospective case-control study (from 2009 to 2012, up to 3 years)
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | PUD in Chronic Hepatitis | No PUD in Lchronic Hepatitis
Number analyzed (Participants) | 13 | 114
mmHg | 3.7 [2.15 to 5.3] | 3.4 [2 to 5.78]

ADVERSE EVENTS:
Arm/Group | Patients With Chronic Hepatitis | Patients With Liver Cirrhosis
Serious Adverse Events (participants affected / at risk) | 0/127 | 0/328
Other Adverse Events (participants affected / at risk) | 0/127 | 0/328

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No